CLINICAL TRIAL: NCT02496312
Title: Quantitative Evaluation of Apathy Close to Real Life Situation by Means of a Multimodal Sensor System Integrated in Healthy Subjects and Patients With Frontotemporal Dementia. Pilot Phase.
Brief Title: Quantitative Evaluation of Apathy Close to Real Life Situation by Means of a Multimodal Sensor System Integrated.
Acronym: ECOCAPTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C15-14; 2015-A0087-42 (Registry Identifier: RCB)
Record Dates: First submitted 2015-07-02; First posted 2015-07-14 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2017-10

CONDITIONS: Apathy; Behavior; Frontotemporal Dementia
Keywords: Apathy; Goal-directed behavior; Quantitative evaluation; Sensor; Ethogram
MeSH Terms: conditions — Lethargy; Behavior; Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ECOCAPTURE (Experimental): Quantitative Evaluation of Apathy Close to Real Life Situation by Means of a Multimodal Sensor System Integrated.
  Interventions: Behavioral: Evaluation of Apathy Close to Real Life Situation

INTERVENTIONS:
Behavioral: Evaluation of Apathy Close to Real Life Situation — Quantitative Evaluation of Apathy Close to Real Life Situation by Means of a Multimodal Sensor System Integrated.

SUMMARY:
The purpose of this study is to provide relevant quantitative evaluation of apathy close to real life situation by means of a multimodal sensor system integrated.

DETAILED DESCRIPTION:
The investigators try to measure the amount of goal-directed behaviour and to detect the pattern of apathy. The main objective of this pilot phase is to select the variables of goal-directed behaviour from the list of metrics providing by the multimodal acquisition system in healthy subjects and patients with frontotemporal dementia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Frontotemporal Dementia (FTD) according to diagnostic criteria reported by Rascovsky et al. (2011).
* Understanding of the instructions and capacity to realize the cognitive tasks.
* Capacity to read, to understand and to sign legal document of information
* Capacity for informed consent for research, capacity to sign consent
* MMSE score > 20
* Absence of other cerebral pathology.
* Absence of psychiatric disease interfering with the assessment of the tests
* Absence of excessive psychotropic use
* Access to National Healthcare Insurance
* Accompanied with a caregiver

Exclusion Criteria:

* Excessive psychotropic use
* Incapacity or refusal to realize the experimental tasks
* Subject deprived of freedom by an administrative or court order
* Subject under legal protective measure.
* Incapacity for informed consent for research
* Participation in another biomedical research
* Airway obstruction risk
* Reduction of activity not attributable to another chronic pathological condition

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2015-10-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of each behavior from the ethogram | 45 min
  [Provided by the video recording and The Observer NOLDUS software]
Frequency of each behavior from the ethogram | 45 min
  [Provided by the video recording and The Observer NOLDUS software]
Duration of each behavior from the ethogram | 45 mn
  [Provided by the video recording and The Observer NOLDUS software]
Number of different behaviors | 45 mn
  [Provided by the video recording and The Observer NOLDUS software]
Activity classes | 45 mn
  [Provided by the MOVE MOVISENS sensor] lying, sitting, ...
Body positions | 45 mn
  [Provided by the MOVE MOVISENS sensor] lying left, ...
Energy expenditure | 45 mn
  [Provided by the MOVE MOVISENS sensor] kcal.
MET | 45 mn
  [Provided by the MOVE MOVISENS sensor] The Metabolic Equivalent of Task. MET level.
Steps | 45 mn
  [Provided by the MOVE MOVISENS sensor] Counting steps.
Activity intensity | 45 mn
  [Provided by the MOVE MOVISENS sensor] g.

CONTACTS AND LOCATIONS:
Overall Officials: Richard LEVY, PhD, MD, Principal Investigator — INSERM UMR_S 1127, ICM

REFERENCES:
- [Background] Robert PH, Clairet S, Benoit M, Koutaich J, Bertogliati C, Tible O, Caci H, Borg M, Brocker P, Bedoucha P. The apathy inventory: assessment of apathy and awareness in Alzheimer's disease, Parkinson's disease and mild cognitive impairment. Int J Geriatr Psychiatry. 2002 Dec;17(12):1099-105. doi: 10.1002/gps.755. PMID 12461757
- [Background] Pasquier F, Lebert F, Lavenu I, Guillaume B. The clinical picture of frontotemporal dementia: diagnosis and follow-up. Dement Geriatr Cogn Disord. 1999;10 Suppl 1:10-4. doi: 10.1159/000051206. PMID 10436334
- [Background] Mayo NE, Fellows LK, Scott SC, Cameron J, Wood-Dauphinee S. A longitudinal view of apathy and its impact after stroke. Stroke. 2009 Oct;40(10):3299-307. doi: 10.1161/STROKEAHA.109.554410. Epub 2009 Aug 27. PMID 19713543
- [Background] Winograd-Gurvich C, Fitzgerald PB, Georgiou-Karistianis N, Bradshaw JL, White OB. Negative symptoms: A review of schizophrenia, melancholic depression and Parkinson's disease. Brain Res Bull. 2006 Oct 16;70(4-6):312-21. doi: 10.1016/j.brainresbull.2006.06.007. Epub 2006 Jul 5. PMID 17027767
- [Background] Marin RS, Firinciogullari S, Biedrzycki RC. Group differences in the relationship between apathy and depression. J Nerv Ment Dis. 1994 Apr;182(4):235-9. doi: 10.1097/00005053-199404000-00008. PMID 10678322
- [Background] Dujardin K, Sockeel P, Delliaux M, Destee A, Defebvre L. The Lille Apathy Rating Scale: validation of a caregiver-based version. Mov Disord. 2008 Apr 30;23(6):845-9. doi: 10.1002/mds.21968. PMID 18307266
- [Background] Lane-Brown AT, Tate RL. Apathy after acquired brain impairment: a systematic review of non-pharmacological interventions. Neuropsychol Rehabil. 2009 Aug;19(4):481-516. doi: 10.1080/09602010902949207. PMID 19533496
- [Background] Czernecki V, Pillon B, Houeto JL, Welter ML, Mesnage V, Agid Y, Dubois B. Does bilateral stimulation of the subthalamic nucleus aggravate apathy in Parkinson's disease? J Neurol Neurosurg Psychiatry. 2005 Jun;76(6):775-9. doi: 10.1136/jnnp.2003.033258. PMID 15897497
- [Background] Le Jeune F, Drapier D, Bourguignon A, Peron J, Mesbah H, Drapier S, Sauleau P, Haegelen C, Travers D, Garin E, Malbert CH, Millet B, Verin M. Subthalamic nucleus stimulation in Parkinson disease induces apathy: a PET study. Neurology. 2009 Nov 24;73(21):1746-51. doi: 10.1212/WNL.0b013e3181c34b34. PMID 19933975
- [Background] Marin RS. Apathy: a neuropsychiatric syndrome. J Neuropsychiatry Clin Neurosci. 1991 Summer;3(3):243-54. doi: 10.1176/jnp.3.3.243. PMID 1821241
- [Background] Levy R, Dubois B. Apathy and the functional anatomy of the prefrontal cortex-basal ganglia circuits. Cereb Cortex. 2006 Jul;16(7):916-28. doi: 10.1093/cercor/bhj043. Epub 2005 Oct 5. PMID 16207933
- [Background] Levy R, Czernecki V. Apathy and the basal ganglia. J Neurol. 2006 Dec;253 Suppl 7:VII54-61. doi: 10.1007/s00415-006-7012-5. PMID 17131230
- [Background] Brown RG, Pluck G. Negative symptoms: the 'pathology' of motivation and goal-directed behaviour. Trends Neurosci. 2000 Sep;23(9):412-7. doi: 10.1016/s0166-2236(00)01626-x. PMID 10941190
- [Background] Muller U, Czymmek J, Thone-Otto A, Von Cramon DY. Reduced daytime activity in patients with acquired brain damage and apathy: a study with ambulatory actigraphy. Brain Inj. 2006 Feb;20(2):157-60. doi: 10.1080/02699050500443467. PMID 16421064
- [Background] Funkiewiez A, Bertoux M, de Souza LC, Levy R, Dubois B. The SEA (Social cognition and Emotional Assessment): a clinical neuropsychological tool for early diagnosis of frontal variant of frontotemporal lobar degeneration. Neuropsychology. 2012 Jan;26(1):81-90. doi: 10.1037/a0025318. Epub 2011 Sep 5. PMID 21895376
- [Result] Batrancourt B, Lecouturier K, Ferrand-Verdejo J, Guillemot V, Azuar C, Bendetowicz D, Migliaccio R, Rametti-Lacroux A, Dubois B, Levy R. Exploration Deficits Under Ecological Conditions as a Marker of Apathy in Frontotemporal Dementia. Front Neurol. 2019 Aug 28;10:941. doi: 10.3389/fneur.2019.00941. eCollection 2019. PMID 31551908
- [Result] Tanguy D, Rametti-Lacroux A, Bouzigues A, Saracino D, Le Ber I, Godefroy V, Morandi X, Jannin P, Levy R, Batrancourt B, Migliaccio R; ECOCAPTURE Study Group. Behavioural disinhibition in frontotemporal dementia investigated within an ecological framework. Cortex. 2023 Mar;160:152-166. doi: 10.1016/j.cortex.2022.11.013. Epub 2022 Dec 28. PMID 36658040
- [Result] Godefroy V, Batrancourt B, Charron S, Bouzigues A, Bendetowicz D, Carle G, Rametti-Lacroux A, Bombois S, Cognat E, Migliaccio R, Levy R. Functional connectivity correlates of reduced goal-directed behaviors in behavioural variant frontotemporal dementia. Brain Struct Funct. 2022 Dec;227(9):2971-2989. doi: 10.1007/s00429-022-02519-5. Epub 2022 Jun 25. PMID 35751676
- [Result] Godefroy V, Batrancourt B, Charron S, Bouzigues A, Sezer I, Bendetowicz D, Carle G, Rametti-Lacroux A, Bombois S, Cognat E, Migliaccio R, Levy R. Disentangling Clinical Profiles of Apathy in Behavioral Variant Frontotemporal Dementia. J Alzheimers Dis. 2022;90(2):639-654. doi: 10.3233/JAD-220370. PMID 36155506